CLINICAL TRIAL: NCT05863676
Title: Ovarian Tissue Cryopreservation in the Setting of Gender-affirming Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Other Study IDs: STUDY19060046
Record Dates: First submitted 2023-04-13; First posted 2023-05-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Gender Dysphoria; Transgender
Keywords: Fertility; Fertility Preservation; Infertility; Gender Affirming; Gender Diverse; Non-Binary; Ovary
MeSH Terms: conditions — Gender Dysphoria; Infertility | interventions — Ovariectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ovarian Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cryopreservation: Participants will have their gonadal tissue cryopreserved.
  Interventions: Procedure: Oophorectomy; Diagnostic Test: Infectious Disease Testing

INTERVENTIONS:
Procedure: Oophorectomy — Ovary will be removed for fertility preservation.
Diagnostic Test: Infectious Disease Testing — Infectious Disease Testing will be done on participants.

SUMMARY:
The goal of this study is to learn about fertility preservation in the gender-diverse community. The main objectives it aims to understand are to:

1. To optimize techniques for cryopreservation of ovarian tissues, including determining efficacy of cryopreservation techniques.
2. To investigate factors affecting ovarian tissue and follicles, such as previous treatment with leuprolide acetate, or hormone therapy

DETAILED DESCRIPTION:
Fertility preservation is an important aspect of care for all patients who may have their fertility compromised secondary to disease, medical treatments, age or other circumstances, including treatments for gender dysphoria. An increasing number of transgender male patients (transitioning female to male) are presenting to fertility clinics for fertility preservation. Studies indicate that parenthood is important for this patient population . Therefore, both the Endocrine Society and the World Professional Association for Transgender Health (WPATH) recommend that fertility preservation be discussed with all patients prior to initiation of medical treatments for gender dysphoria.

For transgender male patients, medical treatment is primarily comprised of testosterone, which is often preceded by GnRH agonists (such as leuprolide acetate) to reduce endogenous estrogen production. There are theoretical concerns about the effects of long-standing hormonal treatment on the gonads and future fertility potential. Regardless of the timing of initiation of GnRH agonist and/or testosterone therapy, fertility preservation counseling is an essential aspect of their care. Egg preservation does require the individual to undergo their natal puberty, and for many trans-males, this is undesirable and even contra-indicated from mental health standpoint, as the suicide rate for transgender youth is 10-times the national average. Ovarian tissue cryopreservation is an alternative option for transgender male patients who desire pubertal blockade and testosterone but have not yet gone through female puberty and are therefore not producing mature eggs.

ELIGIBILITY:
Inclusion Criteria:Two Categories of participants will be eligible for this study.

Category 1 participants must have all criteria listed below:

* Patient with ovaries over the age of 9
* Diagnosed with gender dysphoria; currently on or imminently planning to start gender affirming treatment (hormone blockers or gender-affirming hormones)
* Have a clinical referral for fertility preservation from their primary care physician
* Unwilling to undergo natal puberty or, for patients who have gone through puberty, unwilling to discontinue hormone suppression and/or hormone replacement therapy.

Category 2 participants only fall into this category if they are undergoing gender-affirming surgery. They must have all criteria listed below:

* Patient is 18+ years old
* Diagnosed with gender dysphoria
* Unwilling to undergo natal puberty, or for patients who have gone through puberty, be unwilling to discontinue hormone suppression and/or sex steroid (estrogen) therapy.
* Will be undergoing gender affirming surgery that involves removal of the ovaries.

Exclusion Criteria:

* Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
* Diagnosed with an underlying medical condition that significantly increases their risk of complications from anesthesia and surgery.

Min Age: 9 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients who will undergo gender-affirming treatments and for whom standard of care fertility preservation procedures are not available.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
To optimize techniques for cryopreservation of ovarian tissues, including determining efficacy of cryopreservation techniques. | [10 years]
  Without undergoing puberty in one's natal sex, there are no standard of care fertility preservation options available for these patients. The study will aim to optimize techniques for cryopreservation of ovarian tissues by utilizing the best scientific standards for cryopreservation.
To investigate factors affecting ovarian tissue and follicles, such as previous treatment with leuprolide acetate, or hormone therapy. | [10 years]
  For transgender male patients, medical treatment is primarily comprised of testosterone, which is often preceded by GnRH agonists (such as leuprolide acetate) to reduce endogenous estrogen production. There are theoretical concerns about the effects of long-standing hormonal treatment on the gonads and future fertility potential. The study aims to determine whether factors such as gender-affirming treatment affects the ovarian tissue and follicles by examining tissue donated to research.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh/ University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The Investigators will publish individual participant data. The investigators will also report each individual participants data back to them. Participants will be identified with unique ID numbers. No identifiable information will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: We will share IPD with the patient (and only the patient) within one year of enrollment. We share study protocol ICF with collaborating sites upon request. De-identified IDP is shared with collaborating sites annually.
Access Criteria: De-identified research data will be shared with collaborators via e-mail, and with the broader scientific community via publication and presentations at national/international meetings.